CLINICAL TRIAL: NCT04521010
Title: Staff Absenteeism and Delivery of Healthcare Services During the COVID-19 Pandemic at Wiktor Dega Orthopedic and Rehabilitation Clinical Hospital in Poznań
Brief Title: Staff Absenteeism and Delivery of Healthcare Services During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 3/2020/Reh
Record Dates: First submitted 2020-08-13; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: COVID-19 Pandemic
Keywords: Staff absenteeism; healthcare services
MeSH Terms: conditions — COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Staff absenteeism: A retrospective analysis of above-mentioned data, covering the period January-April 2019 and January-April 2020, was carried out. The evaluation of the staff's absence included all workers employed under an employment contract: 713 workers in 2019 and 747 workers in 2020.
  Interventions: Other: COVID-19 pandemic
- healthcare services: The variable number of employees was a result of the employment dynamics in the subsequent 2 years, due to variable quantity of healthcare services that were contracted with the national payer and changes in the form of employment of some hospital workers
  Interventions: Other: COVID-19 pandemic

INTERVENTIONS:
Other: COVID-19 pandemic — The aim of the study was to evaluate the staff absenteeism in the initial period of the COVID-19 pandemic at Wiktor Dega Orthopedic and Rehabilitation Clinical Hospital in Poznań Poznań as well as to assess the level of performance of medical services that were assigned to the Hospital under contract with National Health Fund, the payer of public health services in Poland.

SUMMARY:
Work attendance of more than 700 hospital workers was evaluated. The assessment of the number of medical services that were performed was based on monthly reports prepared for the national payer of health services.

DETAILED DESCRIPTION:
A retrospective analysis of above-mentioned data, covering the period January-April 2019 and January-April 2020, was carried out. The evaluation of the staff's absence included all workers employed under an employment contract: 713 workers in 2019 and 747 workers in 2020. The variable number of employees was a result of the employment dynamics in the subsequent 2 years, due to variable quantity of healthcare services that were contracted with the national payer and changes in the form of employment of some hospital workers.Three types of analyses were carried out: global analysis, analysis taking into account division into specific professions and the analysis of absence in different hospital organizational units/areas. The absences due to medical reasons, holidays or childcare were analyzed together. The analysis of performing the contracted tasks was shown in relative values ( %). The analysis included the structure of contracted services dividing them into: Orthopedics (alloplasty and others), rehabilitation (person-day), rheumatology (drug trials and others). Considering the rehabilitation unit, it was subdivided into inpatient and outpatient wards due to temporary closure of the outpatient ward.

ELIGIBILITY:
Inclusion Criteria:

all workers employed under an employment contract Exclusion Criteria: not applicable

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 713 workers in 2019 and 747 workers in 2020.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Number of days an individual person was absent | March and April 2019
  Number of days an individual person was absent during period of March and April 2019 (61 days)

OTHER OUTCOMES:
Number of days an individual person was absent | March and April 2020
  Number of days an individual person was absent during period of March and April 2020 (61 days)

CONTACTS AND LOCATIONS:
Overall Officials: Ewa Chlebuś, MD, Principal Investigator — Department of Rehabilitation and Physiotherapy Rehabilitation
Locations (1):
- Department of Rehabilitation and Physiotherapy Rehabilitation,, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No